CLINICAL TRIAL: NCT04334551
Title: A Pilot, Prospective, Non-randomized Study to Evaluate the Safety and Efficacy of Switches From Etravirine to Doravirine, in Experienced Patients With Multiple Class Resistance Including NNRTI Resistance
Brief Title: HIV Switch Trial in Experienced Patients With Multiple Class Resistance Including NNRTI Resistance
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinique du Quartier Latin (Network)
Collaborators: Merck Frosst Canada Ltd. (Industry)
Responsible Party: Principal Investigator, Benoit Trottier, Dr Benoit Trottier Principal Investigator, Clinique du Quartier Latin
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Doravirine and HIV VT#59184
Record Dates: First submitted 2020-03-23; First posted 2020-04-06 (Actual); Last update posted 2021-01-29 (Actual); Status verified 2021-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — doravirine

STUDY DESIGN:
Intervention Model Description: A pilot, prospective, non-randomized study to evaluate the safety and efficacy of switches from etravirine to doravirine, in experienced patients with multiple class resistance including NNRTI resistance
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- switch from etravirine to doravirine (Experimental): switches to doravirine,
  Interventions: Drug: Doravirine

INTERVENTIONS:
Drug: Doravirine — switches from etravirine to doravirine, in experienced HIV patients

SUMMARY:
This is a pilot, open, prospective, non-randomized study to evaluate the safety and efficacy of switches from etravirine to doravirine, in experienced patients with multiple class resistance including NNRTI resistance. The other ARV medication (protease inhibitor, entry inhibitor and integrase inhibitor) that some patients receive, in addition to the NRTI and NNRTI, will not be changed.

The study will be performed only on two sites

DETAILED DESCRIPTION:
The duration of the study will be of 120 weeks: 24 for recruitment and 96 weeks of follow-up. The reasons for the study duration of 2 years is that, up to now, doravirine has not been studied in 2 or 3 classes multi-drug-resistance (MDR) and thus, demonstration of durability of effect over a prolonged period of time is as important as the short-term efficacy.

ELIGIBILITY:
Inclusion Criteria:

- Adult (18 Y.O. or more) women and men infected with HIV.

* Treated with etravirine and at least 2 others ARV in the other classes: NRTI, PI, INSTI, EI, for at least 12 months.
* Virologically controlled (HIV-1 RNA < 50 copies/mL) since at least 6 months. Blips (HIV-ARN ≥ 50 copies/mL, one time, with return to virologic control at the next visit) are allowed.
* Presence of at least one major NNRTI mutation.
* No limitation on the number of previous regimens.
* HCV and HBV-infected patients are allowed

Exclusion Criteria:

High level of resistance to doravirine according to historical resistance tests.

* Level of resistance to doravirine superior to that of etravirine
* Opportunistic or serious active infection or disease
* Active and untreated malignancy.
* Current psychiatric or neurocognitive condition judged by the Investigator to potentially interfere with study visits and procedures
* Pregnancy.
* Active treatment for hepatitis C is forbidden at entry but will be allowed after 3

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2022-07-14 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Percentage of subjects who maintain virologic control . | 24 weeks
  Virologic control is defined by measurement of HIV-1 RNA < 50 copies/mL.

CONTACTS AND LOCATIONS:
Locations (2):
- Clinique Du Quartier Latin, Montreal, Quebec, Canada
- CHU Martinique, Fort-de-France, Fort de France, Martinique

IPD SHARING:
Plan to Share IPD: No